CLINICAL TRIAL: NCT01281969
Title: A Placebo-Controlled Trial of Intravenous Immunoglobulin (IVIG) for PANDAS (Pediatric Autoimmune Neuropsychiatric Disorders Associated With Streptococcal Infections)
Brief Title: Intravenous Immunoglobulin for PANDAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 110058; 11-M-0058 (Other: National Institute of Mental Health)
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2018-08

CONDITIONS: Obsessive-Compulsive Disorder; Children; Anxiety Disorder; Autoimmune Disease; PANDAS
Keywords: Placebo Controlled; Obsessive-Compulsive Disorder; Children and Adolescents; Intravenous Immunoglobulin; PANDAS
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders; Autoimmune Diseases; Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Group A (Experimental): Drug: Gamunex Intravenous Immunoglobulin 2.0 gm/kg total, IV (in the vein), over 2 days
  Interventions: Drug: Gamunex Intravenous Immunoglobulin
- Group B (Placebo Comparator): Drug: Placebo Normal saline, IV (in the vein), over 2 day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gamunex Intravenous Immunoglobulin — 2.0 gm/kg total, IV (in the vein), over 2 days
  Arms: Group A
Drug: Placebo — Normal saline, IV (in the vein), over 2 days
  Arms: Group B

SUMMARY:
Background:

- Some children experience a sudden onset of symptoms similar to those found in obsessive-compulsive disorder that may be caused by the body s reaction to an infection with streptococcal bacteria, most commonly seen as strep throat or scarlet fever. When the body s immune system reacts against brain cells following a streptococcal infection, the condition is known as PANDAS (pediatric autoimmune neuropsychiatric disorders associated with streptococcal infections). The immune system response can be inactivated by treatment with a drug known as intravenous immunoglobulin (IVIG). Because there is insufficient research on IVIG s effects on the immune system of children with PANDAS, including whether IVIG is helpful in treating obsessive-compulsive symptoms related to PANDAS, researchers are interested in examining whether IVIG is an appropriate treatment for PANDAS and its associated symptoms.

Objectives:

- To test the safety and effectiveness of intravenous immunoglobulin for the treatment of obsessive-compulsive disorder in children with PANDAS (pediatric autoimmune neuropsychiatric disorder associated with streptococcal infection).

Eligibility:

- Children between 4 and 12 years of age who have obsessive-compulsive disorder (with or without a tic disorder) with sudden onset of symptoms following Group A streptococcal bacterial infections.

Design:

* Participants will be screened by telephone to obtain medical history and other information, followed by in-person screening at the National Institutes of Health Clinical Center.
* Participants will be admitted to the hospital to receive 2 days of infusions of either IVIG or a placebo. Frequent blood samples, imaging studies, and other tests will be performed during this visit.
* Six weeks after the inpatient stay, participants will return for further blood samples and other tests. Participants who did not receive the study drug, or who received the drug but did not respond to the initial IVIG infusion, will have the option to receive IVIG at this time.
* Followup visits will take place 3 months and 6 months after the first evaluation, followed by yearly follow-ups for 5 additional years.

DETAILED DESCRIPTION:
Objective:

This study is designed to test the safety and efficacy of intravenous immunoglobulin (IVIG) for the treatment of obsessive-compulsive disorder (OCD) symptoms in children with PANDAS (pediatric autoimmune neuropsychiatric disorder associated with streptococcal infection).

Study Population:

Thirty-two male and female children with severe obsessive-compulsive symptoms related to a new onset or first recurrence of symptoms consistent with the PANDAS subtype of OCD.

Design:

his is a multi-site double-blind placebo-controlled trial. Potential subjects will be screened in person at NIMH, and there will be remote video corroboration by a team of collaborators at Yale University. Eligible subjects will be admitted to the 1NW pediatrics inpatient unit at the Clinical Center for further assessment, randomization, and study drug administration according to protocol. Subjects who fail to improve 6 weeks after blinded IVIG/placebo administration (1.0 gm/kg/day of IVIG on two consecutive days; total dose 2.0 gm/kg) will be eligible to receive open-label IVIG.

Outcome Measures:

* Primary: Improvement in obsessions, compulsions, and other neuropsychiatric symptoms.
* Exploratory:

  * Reduction of titers of cross-reactive antibodies (Abs)
  * Resolution of basal ganglia inflammation (as measured by pre-/post-changes in MRI volumetric scans and inflammatory sequences)
  * Normalization of selected serum and CSF cytokines

ELIGIBILITY:
* INCLUSION CRITERIA:

Male and female children 4-13 years of age.

Presence of (Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision) DSM-IV TR OCD with or without a tic disorder.

Moderate or greater severity of symptoms, with a score of greater than or equal to 20 on the Children s Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) and greater than or equal to 4 on the Clinical Global Impression Severity scale (CGI-S).

The acute onset within the previous six months of symptoms in a child previously well, or the first acute recurrence within the previous six months, after a period of relatively complete remission of symptoms. The acuity of symptom onset/exacerbation is key and must be severe, dramatic in onset, and proceed from no/minimal symptoms to maximum severity within 24-48 hours.

Symptom onset or first exacerbation preceded within four months by a GAS infection, as documented by positive throat culture, exposure to documented GAS infection (in a close contact, such as a sibling sharing a bedroom), and/or documented two-fold rise in one or more anti-GAS antibody titers such as anti-streptolysin O, anti-streptococcal DNAaseB, anti-carbohydrate antibodies and others.

Onset/exacerbation of OCD is accompanied by at least three of the following 7 clinical signs and symptoms. The acuity of the comorbid symptoms must be similar to the OCD symptoms and occur in the same time interval.

1. Markedly increased level of anxiety, particularly new onset of separation anxiety.
2. Emotional lability, irritability, aggressive behavior and/or personality change.
3. Sudden difficulties with concentration or learning.
4. Developmental regression ("baby-talk," temper tantrums; behaviors atypical for actual chronological age).
5. Sleep disorder (insomnia, night terrors, refusal to sleep alone).
6. Handwriting deterioration or other sign of motoric dysfunction (including new onset of motor hyperactivity, or presence of choreiform finger movements).
7. Urinary frequency or increased urge to urinate; daytime or night-time secondary enuresis.

EXCLUSION CRITERIA:

History of rheumatic fever, including Sydenham chorea (the neurologic manifestation).

Presence of symptoms consistent with autism, schizophrenia, or other psychotic disorder (unless psychotic symptoms have onset coincident with the possible PANDAS and are attributed to OCD).

Presence of a neurological disorder other than a tic disorder.

IQ <70. Child subjects need to be able to contribute meaningfully to baseline and follow-up ratings, to report adverse effects, and to assent to participation.

Presence of serious or unstable medical illness or psychiatric or behavioral symptoms that would make participation unsafe or study procedures too difficult to tolerate.

IgA deficiency (<20mg/dL). Intravenous immunoglobulin may contain trace IgA, which may very rarely lead to life-threatening anaphylaxis in IgA-deficient participants with anti-IgA antibodies (Misbah 1993).

Hyperviscosity syndromes, which can increase risks associated with IVIG administration.

Need for live virus vaccine within six months after receiving IVIG (which may be 7.5 months from randomization) since IVIG can interfere with effectiveness of such vaccines. IVIG should not be administered sooner than two weeks after administration of a live virus vaccine, for the same reason.

Taking nephrotoxic drugs. Every concomitant medication will be subject to scrutiny and possible consultation with pediatric safety monitors before randomization to study drug. See below as well.

Recent (less than eight weeks) initiation of cognitive-behavior therapy (CBT).

Recent (less than eight weeks) initiation or change in dosage of psychotropic medication for OCD or tic disorder (e.g., serotonin reuptake inhibitors for OCD, alpha-2 agonists or antipsychotics for tic disorders).

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2018-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Swedo, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ballow M, Berger M, Bonilla FA, Buckley RH, Cunningham-Rundles CH, Fireman P, Kaliner M, Ochs HD, Skoda-Smith S, Sweetser MT, Taki H, Lathia C. Pharmacokinetics and tolerability of a new intravenous immunoglobulin preparation, IGIV-C, 10% (Gamunex, 10%). Vox Sang. 2003 Apr;84(3):202-10. doi: 10.1046/j.1423-0410.2003.00286.x. PMID 12670369
- [Background] Benesch M, Kerbl R, Lackner H, Berghold A, Schwinger W, Triebl-Roth K, Urban C. Low-dose versus high-dose immunoglobulin for primary treatment of acute immune thrombocytopenic purpura in children: results of a prospective, randomized single-center trial. J Pediatr Hematol Oncol. 2003 Oct;25(10):797-800. doi: 10.1097/00043426-200310000-00011. PMID 14528103
- [Background] Berrios X. [Recurrent Sydenham's chorea: a rare manifestation of rheumatic disease]. Rev Med Chil. 1986 Mar;114(3):254-6. No abstract available. Spanish. PMID 3492741
- [Derived] Frick LR, Rapanelli M, Jindachomthong K, Grant P, Leckman JF, Swedo S, Williams K, Pittenger C. Differential binding of antibodies in PANDAS patients to cholinergic interneurons in the striatum. Brain Behav Immun. 2018 Mar;69:304-311. doi: 10.1016/j.bbi.2017.12.004. Epub 2017 Dec 9. PMID 29233751
- [Derived] Williams KA, Swedo SE, Farmer CA, Grantz H, Grant PJ, D'Souza P, Hommer R, Katsovich L, King RA, Leckman JF. Randomized, Controlled Trial of Intravenous Immunoglobulin for Pediatric Autoimmune Neuropsychiatric Disorders Associated With Streptococcal Infections. J Am Acad Child Adolesc Psychiatry. 2016 Oct;55(10):860-867.e2. doi: 10.1016/j.jaac.2016.06.017. Epub 2016 Aug 3. PMID 27663941
- [Derived] Gaughan T, Buckley A, Hommer R, Grant P, Williams K, Leckman JF, Swedo SE. Rapid Eye Movement Sleep Abnormalities in Children with Pediatric Acute-Onset Neuropsychiatric Syndrome (PANS). J Clin Sleep Med. 2016 Jul 15;12(7):1027-32. doi: 10.5664/jcsm.5942. PMID 27166296
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-M-0058.html

RESULTS

PARTICIPANT FLOW:
Groups:
- IVIG: Gamunex Intravenous Immunoglobulin: 2.0 gm/kg total, IV (in the vein), over 2 days
- Screened But Not Randomized: Excluded prior to randomization because child did not meet study entry criteria or child refused consent
Period: Overall Study
Arm/Group | IVIG | Placebo | Screened But Not Randomized
Started | 18 | 18 | 12
Completed | 17 | 18 | 0
Not Completed | 1 | 0 | 12
Not completed — not randomized didn't meet criteria | 0 | 0 | 7
Not completed — AE during LP prior to IVIG admin | 1 | 0 | 3
Not completed — not randomized, child consent not given | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVIG | Placebo | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.99 (2.37) | 9.61 (2.32) | 9.30 (2.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 17 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 14 | 16 | 30
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35
Clinical Global Impressions Severity [Number; unit: participants] — Higher values indicate worse severity. Seven points are possible.
  participants
    Moderate (4) | 2 | 3 | 5
    Marked (5) | 8 | 9 | 17
    Severe (6) | 7 | 4 | 11
    Extreme (7) | 0 | 2 | 2
Children's Yale-Brown Obsessive Compulsive Scale Total [Mean (Standard Deviation); unit: units on a scale] — 40 points possible (i.e., range 0-40). Higher scores are more severe symptoms of OCD.
  units on a scale | 26.47 (5.14) | 28.78 (3.98) | 27.65 (4.66)

OUTCOME MEASURES:

1. Primary Outcome: Children's Yale-Brown Obsessive Compulsive Scale Total Score
Description: Active IVIG will be significantly superior to sham IVIG in reducing OC symptoms and providing global relief of neuropsychiatric symptomatology. Total score is reported as the sum of all items and has a range of 0-40. Higher scores indicate more severe symptoms.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 17 | 18
units on a scale | 20.59 (10.12) | 25.67 (8.65)
Statistical Analysis 1: Comparison: Group A vs Group B; Analysis of covariance model controlling for baseline scores. A priori power calculations based on the Perlmutter et al. study (IVIG effect size 1.2) suggested that a sample size of 16 per group would be sufficient to detect an effect size of 1.0 with 80% power; Test type: Superiority or Other; p = 0.44, ANCOVA — p-value is unadjusted. a priori threshold for statistical significance is .05; F(1,34)=0.62, p=.44; Mean Difference (Final Values) = -1.97, 95% CI 2-sided [-7.1 to 3.15]

2. Secondary Outcome: Clinical Global Impressions Improvement
Description: 1=very much improved, 2=much improved, 3=slightly improved, 4=no change, 5=slightly worse, 6=much worse, 7=very much worse
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 17 | 18
units on a scale | 2.88 (1.20) | 3.53 (1.62)
Statistical Analysis 1: Comparison: Group A vs Group B; The Wilcoxon two-sample test was used to compare CGI-Improvement ratings (an ordinal variable) at week 6. Power calculation was based on CYBOCS as primary outcome; Test type: Superiority or Other; p = .12, Wilcoxon (Mann-Whitney) — p-value is not adjusted; Mean rank sum in the placebo group = 19.92; mean rank sum in the IVIG group = 15.97. Z = -1.18, p=.12

3. Secondary Outcome: Clinical Responder to Treatment
Description: Defined as a CGI-I score of 1 or 2 ("much" or "very much" improved) and a decrease in CY-BOCS of at least 30%
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 17 | 18
participants | 6 | 4
Statistical Analysis 1: Comparison: Group A vs Group B; Chi-squared test was used to compare distribution of responders by randomization group. Power calculation was based on CY-BOCS (primary outcome); Test type: Superiority or Other; p = .40, Chi-squared — p-value is not adjusted for multiple comparisons; X2 = 0.72, p=.40

4. Secondary Outcome: The Degree of Treatment Response is Expected to Correlate With the Percentage Reduction in Antinuclear Antibody Titers Following IVIG Administration.
Description: Non-zero values of antinuclear antibodies are considered "positive" and reflective of an ongoing immune response in the individual. First, the number of participants who were classified at baseline as having "positive" antinuclear antibodies was calculated (see outcome measure data table, which states the number (AKA "count") of participants who had "positive" antinuclear antibodies at baseline). We hypothesized that improvement in the ongoing immune response, and therefore a reduction in antinuclear antibody titers, would mediate the effect of IVIG on OCD symptom improvement. However, because very few participants were classified as "positive" at baseline, it was not appropriate to pursue the original question of whether a decline in antinuclear antibodies (i.e., from "positive" to "negative") was related to symptom improvement.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | IVIG | Placebo
Number analyzed (Participants) | 17 | 18
Participants | 8 | 5

5. Secondary Outcome: The Degree of Treatment Response is Also Expected to Correlate With Decreased Inflammation in Specific Regions of the Brain, as Demonstrated by Changes on MRI
Time Frame: 3 Months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AE data were collected 1 week post-infusion and at 6 weeks post infusion.
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 17/17 | 5/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=17) | Group B (N=18)
Headache (General disorders) | 8 | 3
Sore throat (General disorders) | 1 | 2
Stomach or abdominal discomfort (General disorders) | 3 | 1
Nausea (vomiting) (General disorders) | 4 | 1
Muscle/bone/joint pain (General disorders) | 3 | 2
Tiredness/fatigue (General disorders) | 2 | 1
Anxiety (General disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No